CLINICAL TRIAL: NCT00107718
Title: A Phase II Study of IL-18 in Melanoma Patients
Brief Title: Anti-Tumor Activity Of SB-485232 In Patients With Previously Untreated Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB-485232/006
Record Dates: First submitted 2005-04-07; First posted 2005-04-08 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Melanoma
Keywords: IL-18; treatment naive; Phase 2; melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-485232

SUMMARY:
This Phase II study is designed to evaluate the anti-tumor activity of three dose groups of SB-485232 (0.01, 0.1, and 1.0 mg/kg/day) administered intravenously as a single agent in subjects with previously untreated metastatic melanoma.

ELIGIBILITY:
Inclusion criteria:

* Patients must have melanoma that has spread beyond the original location and has not yet been treated.
* Tissue from the spreading melanoma should have been tested to confirm it is melanoma.

Exclusion criteria:

* Patients having hepatitis or HIV infection.
* Taking corticosteroids.
* Patients with the primary site being occular melanoma or patients with melanoma of the brain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-11-15 (Actual); Primary Completion 2006-05-19 (Actual); Study Completion 2006-05-19 (Actual)

PRIMARY OUTCOMES:
Overall response rate of tumor | Up to 12 months
  Tumor response rate (RR) is defined as the percentage of participants achieving either a complete or partial response. Response was at least one measurable lesion as defined by response evaluation criteria for solid tumors (RECIST) criteria or a cutaneous or subcutaneous lesion of at least 1 centimeter (cm) in diameter in one dimension. A distinction was drawn between responses that are confirmed at a repeat assessment and those that are not. If there were unconfirmed responses, then a sensitivity analysis was performed excluding participants with unconfirmed responses. Analysis was performed by both Investigator and independent review committee (IRC). The results were compared and a confirmatory analysis has been presented.

SECONDARY OUTCOMES:
Number of participants with progression free survival | Up to 12 months
  Progression Free Survival is defined as the time from the start of treatment until the first documented sign of disease progression or death due to any cause, whichever occurred first. For participants who did not progress or die, progression free survival was censored at the time of initiation of alternative anti-cancer therapy or time of last contact, whichever occurred first. The times to progression were summarized using the Kaplan-Meier survival curve.
Response duration of SB-485232 for tumor treatment | Up to 12 months
  Response duration defined as the date criteria for Complete Response (CR) or Partial Response (PR) (whichever occured first) was first met until the date criteria for recurrent or progressive disease was first met or death due to any cause was reported, whichever occured first. Time to response was defined as the date study drug was first dosed until the date criteria for CR or PR (whichever occured first) was first met.
Time to response | Up to 12 months
  Response duration defined as the date criteria for CR or PR (whichever occured first) was first met until the date criteria for recurrent or progressive disease was first met or death due to any cause was reported, whichever occured first. Time to response was defined as the date study drug was first dosed until the date criteria for CR or PR (whichever occured first) was first met.
Number of participants with adverse events (AEs), serious adverse events (SAEs), and death. | Up to 12 months
  An AE is any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect.
Change from Baseline In vital signs [systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), and body temperature(BT)] | Baseline (Day 1) to Day 15 and Day 28 of each cycle
  Vital signs including SBP, DBP, HR and BT were taken at Day 1 to Day 15 and follow up visits of each cycle. Baseline assessment was performed pre-dose on Cycle 1 Day 1.
Number of participants with toxicity grade shift of clinical laboratory parameters over period. | Baselie (Cycle1,Day 1), Day 2, Day 15 and Follow up (28 days after last dose of Cycle 13) of each cycle
  Haematology and Clinical Chemistry together are termed as Clinical Laboratory Parameters.Blood samples were collected at Day 1, Day 2, Day 15 and Follow up of each cycle for assessment of clinical chemistry and haematology parameters. Sodium, Potassium, Chloride, Bicarbonate, Calcium, Glucose, Total protein, Albumin, Lactate dehydrogenase, Uric acid, Phosphorus, Creatinine, Blood urea nitrogen, Total bilirubin, Alkaline phosphatase, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) and Magnesium were analyzed in clinical chemistry. Similarly, Hemoglobin, Hematocrit, Platelet count, Total white blood cell count, Neutrophil count, Lymphocyte count, Monocyte count, Eosinophil count and Basophil count wee analyzed in haematology. Number of participants with shift of grades from Baseline in hematology and clinical chemistry parameters toxicities have been summarized here.
Number of participants with immune response to SB485232 over period. | Day 15 of each cycle
  Immunotherapy for melanoma is based on the premise that the immune system can recognize and attack host tumor cells. This may be achieved by either triggering an immune response or by potentiating an otherwise weak immune response that is capable of recognizing the participant's own tumor. Various dosing schedules and combinations involving IFN-α and interleukin (IL)-2 have been tested. The response rate reported with single agent IL-2, as well as for combinations with Interferon-α, range from a low of 3% (as single agent) to a high of 41% (for the combination), with a small percentage of long term responders. The immune response to SB-485232 was assessed by measuring the anti-SB-485232 levels (total immunoglobulin and immunoglobulin E [IgE]) before starting therapy and at specified time points, throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (12):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lutherville-Timonium, Maryland
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
- Australia (8):
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Douglas, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia